CLINICAL TRIAL: NCT06770595
Title: The Effect of Prenatal Breastfeeding Education Through Clinical Demonstrations for Primiparous Women to Prevent Sore Nipples and Engorgement
Brief Title: Breastfeeding Education Through Clinical Demonstration for Primiparous Women to Prevent Sore Nipples and Engorgement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Eka Nurhayati, Dr. Eka Nurhayati, S.ST., M.K.M, Gadjah Mada University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GadjahMadaU03January2025
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Nipple Infection; Nipple Discharge; Engorgement
Keywords: Demonstration clinic; Education; Sore nipples; Engorgement; Breastfeeding
MeSH Terms: conditions — Galactorrhea; Hyperemia; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): The intervention group is third-trimester pregnant women with 34-35 weeks of gestation who received clinical demonstration education breastfeeding about position and attachment. The clinical demonstration is provided by a lactation counselor.
  Respondents in this group will receive education provided face-to-face with the clinical demonstration of breastfeeding positions and attachment. The education was given twice with a duration of 40 minutes to primigravida mothers aged 34-35 weeks gestation. For outcome measurement, A home visit will be carried out by a lactation counselor and enumerator 2 times, the first home visit in 7 days postpartum and the second home visit in 14 days postpartum, to assess breastfeeding positioning and latching practices, assess the baby's sucking, evaluate nipple pain, sore nipples, and engorgement.
  Interventions: Behavioral: breastfeeding positions and attachment practice.

INTERVENTIONS:
Behavioral: breastfeeding positions and attachment practice. — Breastfeeding clinical demonstration is a method of presentation of skills that shows how a particular procedure is performed in position and attachment breastfeeding. Respondents in this group will receive education provided face-to-face once with a duration of 40 minutes, with the following details: first, 25 minutes of education about breastfeeding position and attachment. In this case, the lactation counselor first explains the correct position and attachment for breastfeeding. Respondents were asked to carry out a practical simulation regarding the correct breastfeeding position and attachment using a doll, in this case, the lactation counselor will assess how the mother is positioned and attached. second, 10 minutes of education about swollen breasts and how to deal with them. third, a 10-minute question and answer session related to the educational material provided.

SUMMARY:
Several studies show that breastfeeding problems in the first days of birth pose a significant obstacle to successful breastfeeding. Among the most common breast problems experienced by mothers are breast abscesses, mastitis, nipple pain and sore nipples, engorgement, and flat or inverted nipples. Treatment for sore nipples and breast engorgement is mostly focused on medication. There is very little research that focuses on the impact of interventions regarding breastfeeding techniques carried out during the antenatal period to prevent sore nipples.

Knowing the effect of breastfeeding position and attachment education through clinical demonstration in third-trimester primigravida pregnant women to prevent sore nipples and engorgement.

This research uses quasi-experiments. The population in this research is a third-trimester pregnant woman in the Kasihan, Pajangan, Sewon, Banguntapan, Pleret, and Jetis Community Health Centers. The number of samples in this study was 100 divided into 2, namely 50 intervention groups and 50 control groups. breastfeeding education will be provided to pregnant women at 34-35 weeks of gestation, as led by a lactation counselor. The first session will take place at a puskesmas (public health center), where mothers will receive an e-booklet, followed by 40 minutes of hands-on clinical skills training for those in the intervention group. A second session will take place two weeks after the first session in the form of a home visit only for those in the intervention group. The outcome of this research is position, attachment, effective sucking, nipple pain, sore nipples, and engorgement. T-test and chi-square will be used to test differences and similarities between study groups.

DETAILED DESCRIPTION:
Several studies show that breastfeeding problems in the first days of birth pose a significant obstacle to successful breastfeeding. Among the most common breast problems experienced by mothers are breast abscesses, mastitis, nipple pain and sore nipples, engorgement, and flat or inverted nipples. Treatment for sore nipples and breast engorgement is mostly focused on medication. There is very little research that focuses on the impact of interventions regarding breastfeeding techniques carried out during the antenatal period to prevent sore nipples. Knowing the effect of breastfeeding position and attachment education through clinical demonstration in third-trimester primigravida pregnant women to prevent sore nipples and engorgement.

This research is an experimental study with a quasi-experimental design, the equivalent-time samples design. The population in this research is a third-trimester pregnant woman in the Kasihan, Pajangan, Sewon, Banguntapan, Pleret, and Jetis Community Health Centers. The sampling method in this research used simple random sampling. The number of samples in this study was 100 divided into 2, namely 50 intervention groups and 50 control groups.

breastfeeding education will be provided to pregnant women at 34-35 weeks of gestation, as led by a lactation counselor. The first session will take place at a puskesmas (public health center), where mothers will receive an e-booklet, followed by 40 minutes of hands-on clinical skills training for those in the intervention group. A second session will take place two weeks after the first session in the form of a home visit only for those in the intervention group.

The selection of respondents was determined based on predetermined inclusion criteria. Next, respondents will be confirmed via WhatsApp so that the enumerator can meet with the respondent to provide an explanation regarding the progress of the research and ask for their willingness to participate in the research by signing an informed consent.

Respondents in the control group did not receive any special intervention. Furthermore, respondents were asked to confirm whether they had given birth in both the intervention group and the control group. A home visit will be carried out by a lactation counselor and enumerator one week postpartum. The first visit to the mother to assess breastfeeding positioning and latching practices, assess the baby's sucking, and evaluate nipple pain, sore nipples, and swollen breasts. The second home visit was carried out at 14 days postpartum to assess breastfeeding positioning and latching practices, assess the baby's sucking, and evaluate nipple pain, sore nipples and swollen breasts.

The outcome of this research is knowledge of breastfeeding techniques, position practice, and latching, evaluating the baby's sucking, nipple pain, sore nipples, and engorgement. T-test and chi-square will be used to test differences and similarities between study groups. Multiple logistic regression was used to analyze the impact of the intervention on tender nipples and swollen breasts to control confounding variables. The intervention effect is expressed as crude odds ratio and adjusted odds ratio, and the associated 95% CI will be obtained from the logistic regression model. The odds ratio was reported along with its 95% CI and was considered significantly significant statistics if the P value is <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Primigravida pregnant women who visited the Kasihan, Pajangan, Sewon, Banguntapan, Pleret, and Jetis health service centers
* Single pregnancy
* Mother has a mobile phone with internet access and can use WhatsApp Application
* Plans to stay for 6 months in the research area
* Willing to participate in the research by signing the informed consent

Exclusion Criteria:

* Presence of congenital orofacial abnormalities (labio-gntao-palatoschisis, etc) that make breastfeeding difficult
* Mother with breast problems (history of implant breast surgery)
* The mother or baby experiences problems during labor or postpartum that may lead to research dropouts

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-26 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Breastfeeding positions practice | at birth to 14 days of postpartum
  Mother's ability to practice breastfeeding positions, ordinal scale, measurement using observational checklist totalling 4 items. The value is the positions is not correct at all (if none of the criteria are met), not good positions (if 1 or 2 criteria fulfilled) and good positions (if 3 or 4 criteria fulfilled)
Breastfeeding attachment practice | at birth to 14 days of postpartum
  Mother's ability to practice breastfeeding attachment, ordinal scale, measurement using observational checklist totalling 4 items. The value is the attachment is not correct at all (if none of the criteria are met), not good attachment (if 1 or 2 criteria fulfilled) and good attachment (if 3 or 4 criteria fulfilled)
Evaluate the baby's sucking while breastfeeding | at birth to 14 days of postpartum
  Evaluation the baby's sucking, nominal scale, measurement using observational checklist. Correct sucking technique was defined as the infant having a wide-open mouth, with the tongue under the areola, and expressing milk from the breast by slow, deep sucks. Faulty technique was defined as superficial nipple sucking.
Evaluate of Sore nipples | at birth to 14 days of postpartum
  Evaluation of sore nipples is measured by using Visuals Analog Score (VAS), ordinal scale. Scale 0 (no pain), scale 1-3 (mild), scale 4-6 (Moderate), scale 7-10 (Severe)
Evaluate Nipple pain | at birth to 14 days of postpartum
  Evaluation of nipple pain is measured by Nipple Trauma Score (NTS), ordinal scale. Score 0 (no microscopically visible skin changes), score 1 (erythema or edema or combination of both), score 2 (superficial damage with or without scab formation on < 25% of the nipple surface), score 3 (superficial damage with or without scab formation on > 25% of the nipple surface), score 4 (partial-thickness wound with or without scab formation on < 25% of the nipple surface), score 5 (partial-thickness wound with or without scab formation on > 25% of the nipple surface).
Evaluate Engorgement | at birth to 14 days of postpartum
  Evaluation engorgement is measured by engorgement scale, ordinal scale. Scale 1 (soft, no change), scale 2 (slight change), scale 3 (firm, non-tender), scale 4 (firm, beginning tenderness), scale 5 (firm, tender), scale 6 (very firm and very tender).

SECONDARY OUTCOMES:
Change in knowledge breastfeed techniques | 36 weeks pregnancy to 38 weeks pregnancy
  Ability to give precise answers to questions regarding breastfeeding, Ordinal scale, measurement using a questionnaire totalling 18 items.
  The value is poor knowledge (0-6), enough knowledge (6-12), good knowledge (13-18). The higher score means a better knowledge about breastfeed techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Prasetya Lestari, M.Kes., Study Director — Alma Ata University
Locations (6):
- Indonesia (6):
  - Kasihan Community Health Centers, Bantul, Special Region of Yogyakarta
  - Sewon Community health centers, Bantul, Special Region of Yogyakarta
  - Pajangan Community Health Centers, Bantul, Special Region of Yogyakarta
  - Jetis community health centers, Bantul, Special Region of Yogyakarta
  - Pleret Community Health Centers, Bantul, Special Region of Yogyakarta
  - Banguntapan community health centers, Bantul, Special Region of Yogyakarta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weigert EM, Giugliani ER, Franca MC, Oliveira LD, Bonilha A, Espirito Santo LC, Kohler CV. [The influence of breastfeeding technique on the frequencies of exclusive breastfeeding and nipple trauma in the first month of lactation]. J Pediatr (Rio J). 2005 Jul-Aug;81(4):310-6. Portuguese. PMID 16106316
- [Result] Bergmann RL, Bergmann KE, von Weizsacker K, Berns M, Henrich W, Dudenhausen JW. Breastfeeding is natural but not always easy: intervention for common medical problems of breastfeeding mothers - a review of the scientific evidence. J Perinat Med. 2014 Jan;42(1):9-18. doi: 10.1515/jpm-2013-0095. PMID 24057589
- [Result] Bhandari N, Bahl R, Mazumdar S, Martines J, Black RE, Bhan MK; Infant Feeding Study Group. Effect of community-based promotion of exclusive breastfeeding on diarrhoeal illness and growth: a cluster randomised controlled trial. Lancet. 2003 Apr 26;361(9367):1418-23. doi: 10.1016/S0140-6736(03)13134-0. PMID 12727395
- [Result] Blair A, Cadwell K, Turner-Maffei C, Brimdyr K. The relationship between positioning, the breastfeeding dynamic, the latching process and pain in breastfeeding mothers with sore nipples. Breastfeed Rev. 2003 Jul;11(2):5-10. PMID 14768311
- [Result] Degefa N, Tariku B, Bancha T, Amana G, Hajo A, Kusse Y, Zerihun E, Aschalew Z. Breast Feeding Practice: Positioning and Attachment during Breast Feeding among Lactating Mothers Visiting Health Facility in Areka Town, Southern Ethiopia. Int J Pediatr. 2019 Apr 7;2019:8969432. doi: 10.1155/2019/8969432. eCollection 2019. PMID 31080479
- [Result] Feenstra MM, Jorgine Kirkeby M, Thygesen M, Danbjorg DB, Kronborg H. Early breastfeeding problems: A mixed method study of mothers' experiences. Sex Reprod Healthc. 2018 Jun;16:167-174. doi: 10.1016/j.srhc.2018.04.003. Epub 2018 Apr 6. PMID 29804762
- [Result] Haggkvist AP, Brantsaeter AL, Grjibovski AM, Helsing E, Meltzer HM, Haugen M. Prevalence of breast-feeding in the Norwegian Mother and Child Cohort Study and health service-related correlates of cessation of full breast-feeding. Public Health Nutr. 2010 Dec;13(12):2076-86. doi: 10.1017/S1368980010001771. Epub 2010 Jun 25. PMID 20576199
- [Result] Kent JC, Ashton E, Hardwick CM, Rowan MK, Chia ES, Fairclough KA, Menon LL, Scott C, Mather-McCaw G, Navarro K, Geddes DT. Nipple Pain in Breastfeeding Mothers: Incidence, Causes and Treatments. Int J Environ Res Public Health. 2015 Sep 29;12(10):12247-63. doi: 10.3390/ijerph121012247. PMID 26426034
- [Result] Safari JG, Kimambo SC, Lwelamira JE. Feeding practices and nutritional status of infants in Morogoro Municipality, Tanzania. Tanzan J Health Res. 2013 Jul;15(3):178-85. doi: 10.4314/thrb.v15i3.5. PMID 26591707
- [Result] Teich AS, Barnett J, Bonuck K. Women's perceptions of breastfeeding barriers in early postpartum period: a qualitative analysis nested in two randomized controlled trials. Breastfeed Med. 2014 Jan-Feb;9(1):9-15. doi: 10.1089/bfm.2013.0063. Epub 2013 Dec 4. PMID 24304033
- [Result] Wagner EA, Chantry CJ, Dewey KG, Nommsen-Rivers LA. Breastfeeding concerns at 3 and 7 days postpartum and feeding status at 2 months. Pediatrics. 2013 Oct;132(4):e865-75. doi: 10.1542/peds.2013-0724. Epub 2013 Sep 23. PMID 24062375
- [Result] Zakarija-Grkovic I, Stewart F. Treatments for breast engorgement during lactation. Cochrane Database Syst Rev. 2020 Sep 18;9(9):CD006946. doi: 10.1002/14651858.CD006946.pub4. PMID 32944940